CLINICAL TRIAL: NCT07329049
Title: The Effect of Inspiratory Muscle Training on Cognitive Functions, Cerebral Oxygenation, and Neurotrophic Factor Level in Patients With Obstructive Sleep Apnea Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Feyza Meraklı, Principal investigator, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025/1362
Record Dates: First submitted 2025-12-12; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Obstructive Sleep Apnea Syndrome (OSAS)
Keywords: obstructive sleep apnea syndrome; cognitive function; brain oxygenation; brain-derived neurotrophic factor
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Other): Individuals will receive standard medical treatment. They will be informed about their illnesses, what they need to do, and what they need to be mindful of. A disease-specific informational brochure and a follow-up form will be provided.
  Interventions: Other: Usual Care
- Placebo IMT group (Sham Comparator): In addition to the control group, individuals will undergo low-resistance IMT at 15% of maximum inspiratory pressure every day for 8 weeks.
  Interventions: Device: Placebo inspiratory muscle training
- IMT Group (Active Comparator): Individuals will undergo IMT for 8 weeks in addition to the control group. Resistance will start at 50% of MIP and be gradually increased to 75%.
  Interventions: Device: inspiratory muscle training

INTERVENTIONS:
Device: inspiratory muscle training — In addition to the control group, IMT will be applied for 8 weeks, 7 days a week, twice a day for 15 minutes (30 breaths/3 sets/1-minute break between sets).The intensity of the training provided in IMT will be gradually increased over the 8 weeks.Before starting the training, patients' mouth pressure (MIP) will be measured and the training workload will be determined. During the first 2 weeks of training, 50% of MIP will be applied as the workload, 60% of MIP during weeks 3 and 4, and 75% of MIP during the last 4 weeks.During weekly face-to-face sessions, patients' new MIP values will be measured to determine the new workload.Patients will be given treatment diaries and asked to mark the sessions they have completed.They will be asked to bring these diaries to the physiotherapist once a week during face-to-face sessions. Additionally, during these sessions, patients' use of the IMT device will be checked, and if any errors are detected, device usage will be re-explained.
  Arms: IMT Group
Device: Placebo inspiratory muscle training — In addition to the control group, inspiratory muscle training at 15% of MIP will be administered twice daily for 15 minutes (30 breaths/3 sets/1-minute rest between sets) for 7 days a week over an 8-week period. Patients will be given treatment diaries and asked to mark their sessions and send these diaries to the physical therapist once a week.
  Arms: Placebo IMT group
Other: Usual Care — Individuals will receive standard medical treatment. They will be informed about their illnesses, what they need to do, and what they need to be mindful of. A disease-specific informational brochure and a follow-up form will be provided.
  Arms: Control Group

SUMMARY:
The aim of this clinical study is to examine the effect of an 8-week training program applied to the respiratory muscles that enable breathing in individuals with obstructive sleep apnea syndrome on cognitive functions, oxygenation of brain tissue, and the brain's healing and adaptation processes. The main questions it aims to answer are:

Does respiratory muscle training applied to individuals with obstructive sleep apnea syndrome have a beneficial effect on cognitive functions? Does respiratory muscle training applied to individuals with obstructive sleep apnea syndrome have a beneficial effect on brain oxygenation? Does respiratory muscle training applied to individuals with obstructive sleep apnea syndrome have a beneficial effect on the brain's healing and adaptation processes? A total of 42 individuals with obstructive sleep apnea syndrome will be included in the study. Researchers will compare the effectiveness of respiratory muscle training on individuals with obstructive sleep apnea syndrome by comparing the respiratory muscle training intervention with placebo (low-intensity respiratory muscle training) and usual care. At the beginning of the study, participants' demographic data will be recorded, they will be assessed, their blood will be drawn, and they will be asked to complete a questionnaire. Participants will be given an information brochure and a weekly follow-up form in addition to the necessary medical treatment.

Participants will receive the necessary medical treatment for 8 weeks, fill out the follow-up form provided every day and send it to the researcher once a week, perform inspiratory muscle training exercises for 8 weeks, and meet face-to-face with the researcher once a week.

The follow-up form will be checked every week. All assessments will be repeated at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with moderate OSA using polysomnography
* Aged 18-60
* Not using non-invasive mechanical ventilation (NIMV)
* General health status is stable (The participant does not have an acute -cardiovascular, respiratory, metabolic, or neurological disease; has not experienced a condition requiring hospitalization in the last three months)
* No mental problems that would interfere with cooperation

Exclusion Criteria:

* History of oropharyngeal surgery
* Presence of any neurological, psychological, or cardiac disease
* BMI ≥40 kg/m²
* Presence of hypothyroidism, uncontrolled hypertension, and diabetes
* Having severe obstructive nasal disease
* Being pregnant
* Having cognitive problems
* Having overlap syndrome
* Using drugs, alcohol, sedatives, and hypnotic medications

Exclusion criteria after the study began:

* Exercise group participants with <75% attendance at training sessions
* Failure to attend sessions for 2 consecutive weeks during the treatment period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Digit Span Test | Baseline and 8 weeks
  A subscale of the WAIS-R, this test aims to measure an individual's level of attention. It is administered in two parts using forward and backward sequencing of numbers. Numbers between 1 and 9 are presented to the individual in a random order, and the individual is asked to repeat them in the same sequence. The test is repeated until the individual correctly repeats the sequence twice in a row or until 12 repetitions are reached. In the evaluation of the test, 2 points are awarded for each correct sequence and 1 point for each sequence with one error. Since there are a total of 12 attempts, even if the individual correctly repeats the sequence twice, 2 points are added for each additional attempt required to reach 12 attempts. The maximum possible score on the test is 24. The test will be administered on the first and last days of treatment.
Montreal Cognitive Assessment Scale | Baseline and 8 weeks
  The Turkish version will be used to assess individuals' cognitive function. This scale, which takes approximately 10 minutes to administer, will be administered face-to-face with individuals. The maximum score that can be obtained on the scale is 30. One point is added for individuals with less than 12 years of education. The cutoff value for the scale has been set at <23. The MBDÖ assesses 8 different cognitive function areas: memory, executive functions, visual construction skills, concentration, language, orientation, calculation, and attention. The first and last days of treatment will be evaluated.
Oktem Verbal Memory Processes Test | Baseline and 8 weeks
  The Turkish adaptation of the Verbal Memory Processes Test, developed by Rey in 1964, was created by Oget Oktem.It assesses verbal memory processes such as auditory-verbal learning, memory recording, recall, and recognition.There is a recognition list with 15 words on the front and 45 words on the back.The target word list on the front is repeated 10 times, and after each repetition, the individual is asked to say the words they have learned, which are recorded, and their score is tallied.This score is the Learning Score Dimension. After a 30-40 minute interval, the individual is asked to recall the target words.The score obtained here is the Spontaneous Recall Dimension score. For words that cannot be recalled, three recognition words consisting of one phonemic and one semantic distractor from the recognition list on the back side will be read, and then the individual will be asked whether the word is found in the target word list.The score obtained is the Recognit Dimension Score.
Stroop Test | Baseline and 8 weeks
  This test measures the ability to inhibit inappropriate responses in executive functions, provides information about selective attention under distracting conditions, and demonstrates frontal lobe functions in the brain.Before starting the test, the person is taught which buttons to press for 4 colors (1=yellow, 2=blue, 3=green, and 4=red).Then, the three-stage test begins: In the first stage, the person must identify the color of 24 colored circles appearing sequentially on the screen and press the correct key.In the second stage, the person must recognize only the color in which 24 neutral words of different colors appear sequentially on the screen and press the correct key.The third stage involves the most demanding task: words with color names written in different colors are displayed in sequence on the screen (for ex., the word "red" may be written in blue).The person is asked to focus on the color in which the word is written, not what the word says, and press the correct button
Functional near-infrared spectroscopy (fNIRS) | Baseline and 8 weeks
  Changes in blood flow in the prefrontal cortex related to executive functions will be assessed using functional near-infrared spectroscopy during a verbal fluency task. During the application, a total of 18 optodes will be placed on the dorsolateral prefrontal cortex (DLPFC). Each source/detector pair will be placed approximately 3 centimeters apart in accordance with the EEG 10-20 system. These optodes will be arranged into 24 channels using a soft neoprene cap. The phonemic verbal fluency test will be administered while the individual is wearing the cap, and data from the measurement during the test will be collected using the fNIRS control box and the connected computer. Thus, while the phonemic verbal fluency test is being administered, changes in the concentration of oxyhemoglobin and deoxyhemoglobin in the prefrontal cortex will be recorded using the fNIRS device.
Verbal fluency test | Baseline and 8 weeks
  This test is used to evaluate various executive functions such as attention, semantic memory, information processing speed, task initiation, complex attention, and inhibition of inappropriate responses. The headset will be placed on the individual's head and the optode placement will be adjusted. Recording will then be performed using fNIRS, and a block design consisting of a total of three blocks for the letters 'K, A, S' will be used during the test. Each block covers a total of 140 seconds, consisting of a 10-second pre-rest period, a 60-second activation period, and a 70-second post-rest period. During the activation period, participants will be asked to generate as many words as possible beginning with a specific initial letter. Words should not be proper nouns, repetitions, or numbers. Digital recordings will be made, and the words spoken, their times of utterance, the number of incorrectly spoken words, and the number of repeated words will be recorded. The phonemic fluency sc
Brain-Derived Neurotrophic Factor | Baseline and 8 weeks
  Blood samples will be collected in biochemistry tubes before the first session and after the final session of the 8-week intervention. After 10 minutes of centrifugation, serum will be obtained and stored at -80°C until analysis. BDNF, a key neurotrophic factor for neuronal survival, differentiation, and synaptic plasticity, will be measured using the Human Free BDNF Quantikine ELISA Kit (R&D Systems). The method is based on a sandwich ELISA principle to quantify serum BDNF levels. Venous blood is allowed to clot for 30-60 minutes, centrifuged at 1500-3000 rpm for 10-15 minutes, and stored at -80°C. Before analysis, samples are thawed and processed according to the kit protocol. After incubation, washing, and substrate steps, absorbance is read at 450 nm, and BDNF concentration is calculated from the standard curve. Duplicate measurements are recommended for reliability.

SECONDARY OUTCOMES:
Respiratory muscle strength | Baseline and 8 weeks
  The maximum inspiratory MIP and MEP of the respiratory muscles will be measured using an oral pressure measurement device. Oral pressure measurement for MIP and MEP is a valid and reliable method for assessing respiratory function according to the ATS/ERS protocol. For MIP measurement, the individual is asked to perform a maximum expiration, followed by a maximum inspiration with a nose clip in place, and to hold this for 1-3 seconds. MIP measurement is performed as 3 repeated measurements with no more than a 10% difference between them. The highest value obtained is recorded. For MEP measurement, the individual is asked to perform a maximum inspiration and then, with a nose clip attached, perform the maximum possible inspiration and hold it for 1-3 seconds. Three measurements are taken, with no more than a 10% difference between them. The highest value measured is recorded. To prevent infection risk, single-use, individual mouthpieces and filters will be used during measurement.
Respiratory muscle endurance | Baseline and 8 weeks
  Respiratory muscle strength index (S-index) and peak inspiratory flow rate (PIF) using the dynamic method will be assessed using the portable POWERbreathe K5 device (POWERbreathe K5, HaB International Ltd, Warwickshire, UK). During two distinct phases of the assessment session, patients will perform at least ten consecutive speed-dependent maneuvers (with 4.5 seconds between inspirations). Baseline, warm-up, and post-warm-up assessments will be performed sequentially. During the evaluations, patients will be verbally encouraged to exert maximum effort. At the end of the test, the average and best strength index and PIF values will be examined.
Respiratory function test | Baseline and 8 weeks
  A spirometry test (using the Cosmed Pony FX device) will be performed and evaluated in accordance with the acceptability criteria of the ERS/ATS. The individual's informations are entered into the spirometer device. After the person's nose is closed with a clip, they are asked to place the mouthpiece of the spirometer so that there is no gap around the corners of their mouth. Participants will be given a few practice runs before the test. The first test will be a forced vital capacity measurement. First, the person is asked to take a strong deep breath. After maximal inspiration, the person is asked to exhale forcefully and rapidly until all the air in their lungs is expelled, for as long as possible, and then take another deep inspiration. The test results will determine the measured, predicted, and % predicted values. To minimize infection risk, single-use, individual mouthpieces and filters will be used.
Increasing Speed Shuttle Walk Test | Baseline and 8 weeks
  This test assesses maximal capacity with symptom limitation. There is a good correlation between the increasing pace shuttle walk test and the KPET. During the test, the individual is asked to walk between two cones placed 10 meters apart at an increasing speed for 12 minutes. Each 10-meter distance is defined as one shuttle. The test continues until the individual's heart rate reaches 85% of the expected maximum heart rate, until they are unable to continue the test due to shortness of breath symptoms, or until they complete the test. The main measurement of the test is the walking distance. The minimum clinically meaningful value of the test has been found to be 48 meters. The first and last days of treatment will be evaluated.
Biochemical analyses: Oxidative Stress | Baseline and 8 weeks
  Blood samples will be collected before the first and after the final session of the 8-week treatment. After centrifugation, serum will be obtained and stored at -80°C until analysis. Total Antioxidant Status (TAS) and Total Oxidant Status (TOS) will be measured using Rel Assay Diagnostics kits. TAS reflects the overall antioxidant capacity, based on suppression of color formation in a Fenton-type reaction, and results are expressed as mmol Trolox equiv/L. TOS measures the total oxidant load through oxidation of Fe²⁺ to Fe³⁺, which forms a purple-red complex with xylenol orange; results are expressed as µmol H₂O₂ equiv/L. For both assays, thawed serum, standards, and reagents are pipetted into microplates, incubated, and absorbance is read at 660 nm (TAS) or 560 nm (TOS). The Oxidative Stress Index (OSI) will be calculated as TOS/TAS × 100.
Daytime Sleepiness Assessment: Epworth Sleepiness Scale (ESS) | Baseline and 8 weeks
  The Turkish version will be used to assess individuals' sleepiness during the day. This scale consists of a total of 8 questions, and the maximum possible score is 24. A score of 0-5 is considered normal, 6-10 is normal but indicates increased daytime sleepiness, 11-12 indicates increased but mild daytime sleepiness, 13-15 indicates increased moderate daytime sleepiness, and 16-24 indicates increased severe daytime sleepiness. The first and last days of treatment will be evaluated.
Sleep quality: Actigraphy | Baseline and 8 weeks
  An actigraph is a small, lightweight, watch-like device that can be worn on the wrist. It is non-invasive and continuously records an individual's movement and activity to determine sleep and wakefulness periods. These devices, which can record activity for varying periods depending on the capacity of their micro-sensors, are used in conjunction with sleep diaries to assess sleep patterns and quality (sleep stages, sleep onset latency, total sleep time, number of nighttime awakenings). In our study, we will use the ActiGraph GT3X-BT, a 3-axis accelerometer. Participants will be asked to wear the actigraphy device on the non-dominant wrist for 3 nights (2 weekdays and 1 weekend day) during sleep and to keep a sleep diary. They will be asked to record the times they put on and take off the device, as well as their bedtime, in their sleep diaries.
Pittsburgh Sleep Quality Index (PSQI) | Baseline and 8 weeks
  The Turkish version will be used to assess individuals' sleep quality over the past month. The questionnaire consists of 24 questions, 19 of which are answered by the person administering the questionnaire, and the other 5 are answered by someone sharing the same room with the respondent, if applicable. These 5 questions are not included in the calculation of the survey score. The questions in the survey assess the individual's sleep quality, habitual sleep efficiency, sleep latency and duration, sleep medication use, sleep disorder, and daytime dysfunction in 7 categories. The questionnaire is scored on a scale of 0-21, and a score greater than 5 indicates poor sleep quality.
Anxiety and depression: Hospital Anxiety and Depression Scale (HADS): | Baseline and 8 weeks
  The Hospital Anxiety and Depression Scale (HADS), developed by Zigmond and Snaith, was used to assess patients' depression and anxiety levels within the hospital. The HADS scale, which has also been validated and tested for reliability in Turkish, consists of a total of 14 items, with 7 questions assessing anxiety and 7 assessing depression. Each question is scored from 0 to 3 according to the answer given, and as the total score increases, the severity of depression and anxiety also increases. Each is evaluated on a scale of 21 points, with a cutoff value of 7 being normal, 8-10 being mild, 11-14 being moderate, and 15 or above being severe.
Fatigue Severity Scale | Baseline and 8 weeks
  The Turkish version will be used to determine the individual's fatigue level over the past week. The scale consists of a total of 9 questions and has a Likert-type scoring system where each question can be scored from 1 to 7. A score of 7 indicates that the individual strongly agrees, while a score of 1 indicates that they strongly disagree. The total score is calculated by dividing the total points by 9. A result of <2.8 indicates no fatigue, while a result of >6.1 indicates severe fatigue.
Quality of life assessment: Functional Outcomes of Sleep Questionnaire (FOSQ) | Baseline and 8 weeks
  The Turkish adaptation will be used to assess the individual's OUAS-specific quality of life. The questionnaire consists of 26 questions, including 7 items assessing attention level, 9 items assessing activity level, 2 items assessing social outcomes, and 8 items assessing overall efficiency. Subgroup scores are calculated between 0 and 4, and the total score that can be obtained from the questionnaire is between 4 and 16. The lower the score, the greater the dysfunction.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng YY, Lin SY, Hsu CY, Fu PK. Respiratory Muscle Training Can Improve Cognition, Lung Function, and Diaphragmatic Thickness Fraction in Male and Non-Obese Patients with Chronic Obstructive Pulmonary Disease: A Prospective Study. J Pers Med. 2022 Mar 16;12(3):475. doi: 10.3390/jpm12030475. PMID 35330474
- [Background] Ferreira L, Tanaka K, Santos-Galduroz RF, Galduroz JC. Respiratory training as strategy to prevent cognitive decline in aging: a randomized controlled trial. Clin Interv Aging. 2015 Mar 20;10:593-603. doi: 10.2147/CIA.S79560. eCollection 2015. PMID 25848235
- [Background] Souza AKF, Dornelas de Andrade A, de Medeiros AIC, de Aguiar MIR, Rocha TDS, Pedrosa RP, de Lima AMJ. Effectiveness of inspiratory muscle training on sleep and functional capacity to exercise in obstructive sleep apnea: a randomized controlled trial. Sleep Breath. 2018 Sep;22(3):631-639. doi: 10.1007/s11325-017-1591-5. Epub 2017 Nov 9. PMID 29124630
- [Background] Nobrega-Junior JCN, Dornelas de Andrade A, de Andrade EAM, Andrade MDA, Ribeiro ASV, Pedrosa RP, Ferreira APL, de Lima AMJ. Inspiratory Muscle Training in the Severity of Obstructive Sleep Apnea, Sleep Quality and Excessive Daytime Sleepiness: A Placebo-Controlled, Randomized Trial. Nat Sci Sleep. 2020 Dec 2;12:1105-1113. doi: 10.2147/NSS.S269360. eCollection 2020. PMID 33293881